CLINICAL TRIAL: NCT01754714
Title: Open-label, Randomized, Parallel-Group, Exploratory Study to Investigate the Effects of Different Doses of S-adenosyl-L-methionine (SAMe) in Subjects With Nonalcoholic Steatohepatitis (NASH) and Non-treated Matched Healthy Volunteers as Control Group
Brief Title: Study to Investigate the Effects of Different Doses of S-adenosyl-L-methionine (SAMe) in Subjects With Nonalcoholic Fatty Liver Disease and Non-treated Matched Healthy Volunteers as Control Group
Acronym: EXPO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M13-397; 2012-000975-18 (EudraCT Number)
Record Dates: First submitted 2012-12-19; First posted 2012-12-21 (Estimated); Results first posted 2016-02-19 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-01

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — S-Adenosylmethionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1000 mg SAMe (S-adenosyl-L-methionine) (Experimental)
  Interventions: Drug: SAMe 1000 mg
- 1500 mg SAMe (Experimental)
  Interventions: Drug: SAMe 1500 mg
- 2000 mg SAMe (Experimental)
  Interventions: Drug: SAMe 2000 mg
- No treatment (No Intervention)

INTERVENTIONS:
Drug: SAMe 1000 mg — 1000 mg dose group: one 500 mg capsule fasting in the morning and one 500 mg capsule before dinner
  Arms: 1000 mg SAMe (S-adenosyl-L-methionine)
Drug: SAMe 1500 mg — 1500 mg dose group: two 500 mg capsules fasting in the morning and one 500 mg capsule before dinner
  Arms: 1500 mg SAMe
Drug: SAMe 2000 mg — 2000 mg dose group: two 500 mg capsules fasting in the morning and two 500 mg capsules before dinner
  Arms: 2000 mg SAMe

SUMMARY:
Investigation the Effects of Different Doses of SAMe in Subjects with Nonalcoholic Fatty Liver Disease and non-treated matched healthy volunteers as control group

ELIGIBILITY:
Inclusion Criteria

* Subjects with non-alcoholic steatohepatitis based on histology in medical history within the last 3 years
* Subjects in a stable metabolic condition since histology for NASH (Non-alcoholic Steatohepatitis)

Exclusion Criteria

* Subjects with extrahepatic biliary obstruction
* Subjects with primary sclerosing cholangitis (PSC)
* Subjects with primary biliary cirrhosis (PBC)
* Any form of malignancy within the past 5 years and/or basal cell carcinoma and squamous cell carcinoma of the skin within the past two years
* History of active substance abuse (oral, inhaled or injected) within one year prior to the study
* Subjects with renal impairment (creatinine level of >2.0 mg/dL)
* Subjects with a known hypersensitivity to the active substance (ademetionine) or methionine or to any of the inactive ingredients
* Subjects with known genetic defects affecting the methionine cycle and/or causing homocystinuria and/or hyperhomocysteinemia (e.g., cystathionine beta-synthase deficiency, Vitamin B12 metabolism defect)
* Subjects on total parenteral nutrition in the year prior to screening
* Subjects after or planned for bariatric surgery (jejunoileal bypass or gastric weight loss surgery)
* Extrahepatic cholestasis (proven by ultrasound)
* Subjects with alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 5 upper limit of normal (ULN)
* Subject with serum total bilirubin (STB) > 5 ULN
* Subjects after liver transplantation and subjects on the waiting list for liver transplantation
* Subjects with any of the following disease in medical history:
* Viral hepatitis (serum positive HBcAb (hepatitis B core antibody) or Hepatitis C Virus (HCV) ribonucleic acid (RNA)
* Evidence of autoimmune liver disease
* Wilson's disease
* Hemochromatosis
* Alpha-1-antitrypsin deficiency
* Known positivity for antibody to human immunodeficiency virus (HIV)
* Known heart failure of New York heart Association class 3 or 4
* Current or history of significant alcohol consumption for a period of more than three consecutive months within five years prior to screening (significant alcohol consumption is defined as > 3 U (unit)/day for men and > 2 U/day for women, on average) or binge drinking or inability to reliably quantify alcohol consumption.
* Clinical or histological evidence of cirrhosis F4
* Subjects with history of biliary diversion
* Subjects with uncontrolled diabetes mellitus defined by HbA1c (hemoglobin A1c) > 8.0 % at screening
* Concomitant medication of B12, folate, betaine or choline
* Concomitant treatment with glitazone within the past year prior to the study
* Subjects with known folate or B12 deficiency
* BMI (body mass index) > 40 kg/m2
* History of major depression diagnostic and statistical manual of mental disorders (DSM-IV) or bipolar disease
* Women of childbearing potential: positive urine pregnancy test during screening or unwillingness to use an effective form of birth control during the study.
* Breastfeeding women
* Any condition that, in the opinion of the investigator, does not justify the patient's inclusion into the study
* Investigational drug intake within one month prior to the study
* Active, serious medical disease with likely life-expectancy less than five years
* Uncooperative attitude or reasonable likelihood for non-compliance with the protocol or any other reason that, in the investigator's opinion, prohibits the inclusion of the subject into the study
* Legal incapacity or limited legal capacity, or who are incarcerated.
* Inability to return for scheduled visits.
* Inability to understand and follow the requirements of the protocol in the local language

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suntje Sander-Struckmeier, PhD, Study Director — Abbott
Locations (32):
- France (8):
  - Site Reference ID 93914, Amiens
  - Site Reference ID 93895, Angers
  - Site Reference ID 93894, Bobigny
  - Site Reference ID 93913, Montpellier
  - Site Reference ID 93916, Nice
  - Site Reference ID 93915, Paris
  - Site Reference ID 93893, Paris
  - Site Reference ID 93896, Pessac
- Germany (9):
  - Site Reference ID 93953, Bonn
  - Site Reference ID 93954, Frankfurt
  - Site Reference ID 93935, Freiburg im Breisgau
  - Site Reference ID 93955, Halle
  - Site Reference ID 93917, Hanover
  - Site Reference ID 93933, Homburg
  - Site Reference ID 94015, Leipzig
  - Site Reference ID 93918, Mainz
  - Site Reference ID 94014, Ulm
- Poland (7):
  - Site reference ID/Investigator # 109455, Bydgoszcz
  - Site Reference ID 93958, Chorzów
  - Site Reference ID 93973, Krakow
  - Site Reference ID 93956, Lodz
  - Site Reference ID 93957, Mysłowice
  - Site Reference ID 93974, Warsaw
  - Site Reference ID 93975, Wroclaw
- Russia (8):
  - Site reference ID ORG-000905, Krasnoyarsk
  - Site reference ID ORG-000906, Moscow
  - Site reference ID ORG-000900, Nizhny Novgorod
  - Site reference ID ORG-000907, Novosibirsk
  - Site reference ID ORG-000903, Omsk
  - Site reference ID ORG-000920, Rostov-on-Don
  - Site reference ID ORG-000904, Samara
  - Site reference ID ORG-000901, Stavropol

RESULTS

PARTICIPANT FLOW:
Groups:
- No Treatment: No study drug was administered
Period: Overall Study
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Started | 27 | 27 | 26 | 28
Completed | 27 | 26 | 24 | 27
Not Completed | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment | Total
Number analyzed (Participants) | 27 | 27 | 26 | 28 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 24 | 23 | 21 | 91
  >=65 years | 4 | 3 | 3 | 7 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (13.8) | 50.0 (12.3) | 49.5 (14.2) | 56.6 (11.6) | 51.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 9 | 11 | 45
  Male | 12 | 17 | 17 | 17 | 63
Region of Enrollment [Number; unit: participants]
  Russian Federation | 5 | 6 | 5 | 2 | 18
  Poland | 3 | 2 | 6 | 6 | 17
  France | 6 | 5 | 4 | 9 | 24
  Germany | 13 | 14 | 11 | 11 | 49

OUTCOME MEASURES:

1. Primary Outcome: Methionine Elimination Half-life Measured in Blood.
Description: After the methionine load, blood samples will be obtained at 0.5, 1, 1.5, 3, 4.5, 6, 7.5 and 9 hours. Plasma will be analyzed for methionine.
Time Frame: 0.5, 1, 1.5, 3, 4.5, 6, 7.5 and 9 hours*at Week 7*
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
hour | 4.29 (1.86) | 4.66 (1.57) | 4.25 (1.64) | 4.26 (1.44)

2. Secondary Outcome: Fasting Methionine Concentration of Average Methionine Concentration Versus Time Curve.
Description: as for outcome 1
Time Frame: 0.5, 1, 1.5, 3, 4.5, 6, 7.5 and 9 hours*at Week 7*
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
mcg/mL | 4.02 (0.92) | 3.81 (0.67) | 5.68 (10.13) | 5.62 (8.53)

3. Secondary Outcome: 13 Carbon (Natural, Stable Isotope of Carbon) Methionine Breath Test
Description: parameters cumulative percentage dose of 13 carbon recovered after 30, 60, 90 minutes (cPDR30, cPDR60, cPDR 90) will be evaluated
Time Frame: 0.5, 1, 1.5, 3, 4.5, 6, 7.5 and 9 hours*at Week 7*
Measure: Mean (Standard Deviation); unit: percentage of recovery
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
percentage of recovery
  13C methionine breath test recovery at 30 min (%) | 0.93 (0.73) | 0.77 (0.51) | 0.88 (0.66) | 0.69 (0.55)
  13C methionine breath test recovery at 60 min (%) | 3.66 (1.99) | 3.49 (1.74) | 3.61 (1.78) | 2.98 (1.72)
  13C methionine breath test recovery at 90 min (%) | 6.69 (2.75) | 6.60 (2.56) | 6.68 (2.48) | 5.74 (2.56)

4. Secondary Outcome: Hepatic Panel (Liver Laboratory Parameters)
Description: Serum Total Bilirubin (STB), Serum Conjugated Bilirubin (SCB), liver-alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), Gamma Glutamyl Transpeptidase (GGT)
Time Frame: change from baseline at 6 weeks
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
U/L
  ALP | 1.9 (7.9) | -0.1 (13.7) | 3.4 (24.1) | -6.0 (16.9)
  ALT | -6.2 (19.5) | -6.3 (23.5) | -4.9 (32.2) | -11.9 (33.4)
  AST | -5.1 (15.7) | -3.0 (16.5) | -1.2 (10.7) | -11.6 (27.7)
  GGT | -1.1 (33.7) | -10.6 (62.7) | -2.7 (35.7) | -12.3 (48.1)

5. Secondary Outcome: Metabolic Panel (Metabolic Laboratory Parameters)
Description: Fasting lipid profile (cholesterol, HDL (High Density Lipoprotein), LDL (Low Density Lipoprotein)), amino acid profile, homeostasis model assessment (HOMA-R) and fasting glucose.
Time Frame: change from baseline at 6 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
mmol/L
  Cholesterol | -0.131 (0.593) | 0.046 (0.921) | -0.265 (0.601) | -0.134 (0.659)
  HDL | -0.094 (0.166) | -0.046 (0.254) | -0.098 (0.169) | -0.075 (0.188)
  LDL | 0.125 (0.452) | 0.182 (0.762) | -0.202 (0.589) | -0.112 (0.558)
  HOMA-R | 0.837 (13.232) | 0.127 (3.763) | -1.549 (13.321) | 3.432 (10.837)
  Glucose | -0.068 (0.968) | 0.490 (1.486) | -0.163 (1.009) | -0.121 (1.610)

6. Other Pre Specified Outcome: Immunological/Anti-oxidant Panel (Immunological and Anti-oxidant Laboratory Parameters)
Description: Cytokine profile ( Interleukin-6, IL-8, IL-10 (IL), Tumor Necrosis Factor (TNF -α), monocyte chemoattractant protein (MCP-1), and Granulocyte-colony stimulating factor (G-CSF ).
Time Frame: change from baseline at 6 weeks
Description (as registered): C-reactive Protein (CRP)
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
pg/mL
  IL-6: n= (27,24,23,27) | 0.0603 (2.0263) | -0.9254 (6.4599) | -1.3194 (4.5779) | 0.1597 (1.6243)
  IL-8: n= (8,6,7,9) | -14.41 (41.07) | 0.65 (13.37) | -78.73 (187.51) | -6.17 (16.94)
  IL-10: n= (1,2,1,2) | 0.270 (NA) — not calculated as there was data of only 1 patient available | -0.045 (0.106) | -0.300 (NA) — not calculated as there was data of only 1 patient available | 1.600 (1.146)
  TNF-alpha: n= (24,24,20,27) | -0.127 (0.414) | -1.083 (4.782) | -0.601 (2.136) | -0.187 (1.114)
  MCP-1: n= (27,25,24,27) | -29.75 (154.75) | -20.60 (79.71) | -40.15 (96.21) | -44.51 (114.85)
  G-CSF: n= (5,4,1,0) | -20.0 (52.8) | -0.5 (9.7) | 20.0 (NA) — not calculated as there was data of only 1 patient available | NA (NA) — not calculated as there was no data of patients available

7. Other Pre Specified Outcome: Fibrosis and Apoptosis Markers (Fibrosis and Apoptosis Laboratory Markers)
Description: Non-invasive test for liver disease (ActiTest)/Fibrotest
  FibroTest® : diagnoses hepatic fibrosis ActiTest® : assesses viral necro-inflammatory activity Scores between 0 and 1, the higher the score the worse
  The FibroTest score is calculated from the results of a six-parameter blood test, combining six serum markers with the age and gender of the patient:Alpha-2-macroglobulin, Haptoglobin, Apolipoprotein A1, Gamma-glutamyl transpeptidase (GGT), Total bilirubin, and Alanine transaminase (ALT). ALT is used in a second assessment called ActiTest that is part of FibroTest.
Time Frame: change from baseline at 6 weeks
Description (as registered): Caspase-cleaved cytokeratin (CK 18)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
scores on a scale
  ActiTest Score | -0.017 (0.098) | -0.022 (0.137) | -0.002 (0.168) | -0.042 (0.096)
  Fibrotest Score | 0.036 (0.097) | 0.028 (0.093) | 0.050 (0.125) | 0.020 (0.068)

8. Secondary Outcome: The Metabolic Clearance Rate Measured in the Blood.
Description: as for outcome 1
Time Frame: 0.5, 1, 1.5, 3, 4.5, 6, 7.5 and 9 hours*at Week 7*
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
L/h | 8.86 (2.93) | 9.83 (3.27) | 10.05 (4.32) | 8.23 (2.30)

9. Secondary Outcome: Methionine Volume of Distribution at Week 7 (L)
Description: After the methionine load, blood samples will be obtained at 0.5, 1, 1.5, 3, 4, 5, 6, 7.5 and 9 hours. Plasma will be analyzed for methionine.
Time Frame: 0.5, 1, 1.5, 3, 4.5, 6, 7.5 and 9 hours*at Week 7*
Measure: Mean (Standard Deviation); unit: L
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
L | 54.40 (18.43) | 62.84 (14.04) | 64.58 (17.77) | 8.23 (53.98)

10. Secondary Outcome: 13 Carbon (Natural, Stable Isotope of Carbon) Methionine Breath Test
Description: Peak
Time Frame: 0.5, 1, 1.5, 3, 4.5, 6, 7.5 and 9 hours*at Week 7*
Measure: Mean (Standard Deviation); unit: Atom %C13
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
Atom %C13 | 1.0972 (0.0062) | 1.0964 (0.0052) | 1.0964 (0.0053) | 1.0949 (0.0045)

11. Secondary Outcome: 13 Carbon (Natural, Stable Isotope of Carbon) Methionine Breath Test
Description: Time to peak
Time Frame: 0.5, 1, 1.5, 3, 4.5, 6, 7.5 and 9 hours*at Week 7*
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
minutes | 70.0 [50.0 to 80.0] | 70.0 [60.0 to 90.0] | 70.0 [50.0 to 80.0] | 70.0 [60.0 to 90.0]

12. Secondary Outcome: Metabolic Panel (Metabolic Laboratory Parameters)
Description: Fasting plasma insulin
Time Frame: Change from baseline at 6 weeks
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
pmol/L | 0.3 (191.0) | -13.6 (115.5) | -13.1 (248) | 69.1 (309.0)

13. Secondary Outcome: Metabolic Panel (Metabolic Laboratory Parameters)
Description: glycosylated hemoglobin (HbA1c)
Time Frame: change from baseline at 6 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
Percentage | -0.08 (0.28) | -0.06 (0.36) | -0.05 (0.32) | 0.02 (0.33)

14. Secondary Outcome: Metabolic Panel (Metabolic Laboratory Parameters)
Description: Adiponectin
Time Frame: change from baseline at 6 weeks
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
mcg/mL | 0.754 (4.191) | 0.425 (1.199) | 0.219 (1.661) | 0.045 (1.515)

15. Secondary Outcome: Immunological/Anti-oxidant Panel (Immunological and Anti-oxidant Laboratory Parameters)
Description: C-reactive Protein (CRP)
Time Frame: change from baseline at 6 weeks
Description (as registered): glutathione in erythrocytes
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
nmol/L | -0.79 (15.51) | -0.80 (14.90) | -8.02 (20.40) | -4.80 (12.8)

16. Secondary Outcome: Immunological/Anti-oxidant Panel (Immunological and Anti-oxidant Laboratory Parameters)
Description: glutathione in erythrocytes
Time Frame: change from baseline at 6 weeks
Description (as registered): oxidative stress marker (isoprostane level)
Measure: Mean (Standard Deviation); unit: mcmol/g
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
mcmol/g | -0.24 (2.06) | -0.21 (1.01) | 0.05 (1.41) | -0.30 (1.33)

17. Secondary Outcome: Immunological/Anti-oxidant Panel (Immunological and Anti-oxidant Laboratory Parameters)
Description: oxidative stress marker (isoprostane level)
Time Frame: change from baseline at 6 weeks
Description (as registered): Cytokine profile ( Interleukin-6, IL-8, IL-10 (IL), Tumor Necrosis Factor (TNF -α), monocyte chemoattractant protein (MCP-1), and Granulocyte-colony stimulating factor (G-CSF ).
Measure: Mean (Standard Deviation); unit: ng/mg Crea
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
ng/mg Crea | -0.223 (0.801) | 0.116 (0.699) | 0.290 (0.691) | -0.223 (0.641)

18. Secondary Outcome: Fibrosis and Apoptosis Markers (Fibrosis and Apoptosis Laboratory Markers)
Description: Caspase-cleaved cytokeratin (CK 18)
Time Frame: change from baseline at 6 weeks
Description (as registered): Hyaluronic acid
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
U/L | -126.8 (401.1) | -136.6 (257.3) | -47.0 (157.3) | -143.2 (532.5)

19. Secondary Outcome: Fibrosis and Apoptosis Markers (Fibrosis and Apoptosis Laboratory Markers)
Description: Hyaluronic acid
Time Frame: change from baseline at 6 weeks
Description (as registered): Non-invasive test for liver disease (ActiTest)/Fibrotest
  FibroTest® : diagnoses hepatic fibrosis ActiTest® : assesses viral necro-inflammatory activity Scores between 0 and 1, the higher the score the worse
  The FibroTest score is calculated from the results of a six-parameter blood test, combining six serum markers with the age and gender of the patient:Alpha-2-macroglobulin, Haptoglobin, Apolipoprotein A1, Gamma-glutamyl transpeptidase (GGT), Total bilirubin, and Alanine transaminase (ALT). ALT is used in a second assessment called ActiTest that is part of FibroTest.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
ng/mL | 4.67 (48.52) | 2.03 (32.26) | 9.40 (59.63) | 3.02 (46.56)

20. Secondary Outcome: Area Under Curve (AUC) of Average Methionine Concentration Versus Time Curve
Description: as for outcome 9
Time Frame: 0.5, 1, 1.5, 3, 4, 5, 6, 7.5 and 9 hours *at Week 7*
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
mcg/mL | 440.09 (149.96) | 399.30 (148.90) | 425.24 (231.88) | 460.57 (135.63)

21. Secondary Outcome: Hepatic Panel (Liver Laboratory Parameters)
Description: ALT/AST ratio
Time Frame: change from baseline at 6 weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Number analyzed (Participants) | 27 | 26 | 24 | 27
Ratio | -0.02 (0.23) | 0.01 (0.21) | 0.03 (0.18) | -0.01 (0.27)

ADVERSE EVENTS:
Arm/Group | 1000 mg SAMe (S-adenosyl-L-methionine) | 1500 mg SAMe | 2000 mg SAMe | No Treatment
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/24 | 1/28
Other Adverse Events (participants affected / at risk) | 7/27 | 4/27 | 7/24 | 2/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1000 mg SAMe (S-adenosyl-L-methionine) (N=27) | 1500 mg SAMe (N=27) | 2000 mg SAMe (N=24) | No Treatment (N=28)
head injury and neck injury before start of treatment (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1000 mg SAMe (S-adenosyl-L-methionine) (N=27) | 1500 mg SAMe (N=27) | 2000 mg SAMe (N=24) | No Treatment (N=28)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No